CLINICAL TRIAL: NCT05587608
Title: US-guided Combined Segmental Thoracic Spinal Epidural Anesthesia in Comparison With General Anesthesia for Upper Abdominal and Breast Surgeries - A Randomized Control Study
Brief Title: US-guided Thoracic Spinal Epidural Anesthesia VS GA for Abdominal and Breast Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Egypt Cancer Institute (Other)
Collaborators: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Ali M. Elzohry, clinical lecturer, South Egypt Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: segmental thoracic TEA-spinal
Record Dates: First submitted 2022-10-14; First posted 2022-10-20 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound-guided thoracic segmental spinal group (Active Comparator): given ultrasound-guided thoracic segmental spinal heavy Marcaine plus 25 ug fentanyl at the level of T10 interlaminar space.
  Interventions: Procedure: combined thoracic segmental spinal epidural anesthesia
- General anesthesia group (No Intervention): General anesthesia (control)

INTERVENTIONS:
Procedure: combined thoracic segmental spinal epidural anesthesia — ultrasound guided thoracic segmental spinal anesthesia at the level of T10 interlaminar space , patients will be in sitting position, spinal needle is then introduced through the epidural needle not more than 0.5 cm beyond the Dura matter. 2cc of heavy Marcaine plus 25 ug fentanyl are injected through the spinal needle.
  Arms: ultrasound-guided thoracic segmental spinal group

SUMMARY:
Ultrasound-guided combined thoracic segmental spinal epidural anesthesia in comparison with general anesthesia in upper abdominal and breast surgery.

DETAILED DESCRIPTION:
The first group (S) will be given ultrasound-guided thoracic segmental spinal anesthesia at the level of T10 interlaminar space, patients will be in sitting position, a combined spinal epidural tray will be used. In this group, SonoSite C60x/5-2 MHz M-Turbo Convex Probe ultrasound Transducer to identify the T10 interlaminar space and after complete sterilization, the investigator will introduce the epidural needle in a Paramedian in plan approach till the epidural space. The spinal needle is then introduced through the epidural needle not more than 0.5 cm beyond the Dura matter. 2cc of heavy Marcaine plus 25 ug fentanyl are injected through the spinal needle. The epidural catheter is then threaded through the Touhy needle after withdrawal of the spinal needle to keep only 4cm up in the epidural space.

ELIGIBILITY:
Inclusion Criteria:

* All upper abdominal and laparoscopic surgeries
* ASA I-III CLASS
* Age between 18 and 60

Exclusion Criteria:

Contraindication of regional ASA More than III Age less than18 or more than 60 Psychological troubles

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2022-10-14 (Actual)

PRIMARY OUTCOMES:
MAP | Change from Baseline Systolic Blood Pressure at one day post operative
  mean arterial pressure

CONTACTS AND LOCATIONS:
Locations (1):
- South Egypt Cancer Institute, Assiut University, Arab Republic of Egypt, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided